CLINICAL TRIAL: NCT02922049
Title: Probe-based Confocal Laser Endomicroscopy in Accurate Histopathologic Diagnosis of Neoplastic Gastrointestinal Lesion
Brief Title: pCLE in the Detection of Esophageal and Gastric Lesions and Intestinal Metaplasia or Dysplasia in Patients After Endoscopic Treatment of BORN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute for Clinical and Experimental Medicine (Other Government)
Responsible Party: Principal Investigator, Doc. (Ass. prof.) Jan Martinek, MD, PhD, AGAF, Ass. Prof. MD. Ph.D. AGAF, Institute for Clinical and Experimental Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16-27648A; G280 (Other: IKEM)
Record Dates: First submitted 2016-09-23; First posted 2016-10-03 (Estimated); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Barrett's Esophagus
Keywords: Probe Based Confocal Laser Endomicroscopy (pCLE); Barrett's esophagus; BORN; Intestinal metaplasia
MeSH Terms: conditions — Barrett Esophagus | interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- pCLE vs. biopsies with histopathology (Other): The investigators will compare diagnostic accuracy and sensitivity of pCLE with standard biopsies in patients with esophageal and gastric lesions and in patients after completed endoscopic treatment of BORN.
  All samples taken by biopsies will be correlated with the images taken by pCLE in the detection of lesions, intestinal metaplasia, dysplasia and buried glands.
  Interventions: Other: Biopsies with histopathology

INTERVENTIONS:
Other: Biopsies with histopathology — All samples taken by biopsies will be correlated with the images taken by CLE.

SUMMARY:
To assess diagnostic accuracy and clinical effectiveness including cost-effectiveness analysis of pCLE in patients after finishing the endoscopic treatment of BORN in detecting persistent/recurrent IM, recurrent neoplasia and buried glands.

DETAILED DESCRIPTION:
Confocal laser endomicroscopy (CLE) has been developed to overcome the limitations of the current endoscopic sampling techniques. CLE allows detailed examination of cellular structures since it provides images very similar to images which a pathologist can see in the microscope. At present, probe based CLE (pCLE) is the only available technology of endomicroscopy. Before optical biopsy, a fluorescein is given intravenously and then fluorescent light coming from a horizontal special focal plane is detected during pCLE of the digestive system.

CLE provide real-time histopathological diagnosis and can lead to an immediate endoscopic treatment in case of early esophageal and gastric neoplasia.

Patients after treatment of Barrett's esophagus related esophageal neoplasia (dysplasia or early cancer) should be surveilled endoscopically with biopsies to rule out relapse of Barrett's esophagus or neoplasia.

Project A - pCLE in the detection of esophageal and gastric lesions:

We plan to investigate the diagnostic accuracy of pCLE (compared to standard histopathology) in patients with endoscopically diagnosed early esophageal and gastric lesions.

Project B - pCLE in the detection of persistent/recurrent intestinal metaplasia/dysplasia in patients after endoscopic treatment of BORN:

Investigators plan to perform a prospective cross-over study comparing the diagnostic accuracy and sensitivity of pCLE with standard biopsies in patients after completed endoscopic treatment of BORN. Surveillance endoscopies are focused on detection of persistent/recurrent IM or dysplasia (ev. neoplasia). BORN is defined as low-grade dysplasia (confirmed by a specialized esophageal pathologist) or as high grade dysplasia or early adenocarcinoma. Investigators will also examine the ability of pCLE to detect buried glands after radiofrequency ablation.

Methods:

Project A:

Patients referred to our department with a suspect and endoscopically visible lesion in the esophagus or stomach will undergo pCLE during a standard upper GI endoscopy with pCLE. After a real-time diagnosis (made by the endoscopist), the standard tissue sampling (biopsies, endoscopic resection or dissection) followed by a standard histopathological tissue assessment will follow.

Project B:

During one of surveillance endoscopies in patients after finishing the endoscopic treatment of BORN (interval depends on baseline diagnosis), pCLE will be performed in the cardia, neo-Z-line, esophagus body and visible lesions, and images will be stored. Thereafter, standard biopsies will be taken and sent for histopathological analysis.

For optical biopsy, endoscopist (real time) and two expert pathologists will independently blindly evaluate each "optical specimen". The standard biopsy specimen will be assessed independently by a pathologist not assessing the optical biopsy. Results of optical biopsy will be compared with results of standard biopsy.

Main hypothesis:

Project A:

pCLE is not inferior to standard biopsy (or resection) specimen in histopathological diagnosing of esophageal/gastric lesions.

Project B:

pCLE is not inferior compared to standard biopsies in detecting persistent/recurrent IM, recurrent neoplasia and buried glands.

ELIGIBILITY:
Inclusion Criteria:

* age > 18
* macroscopic lesion of esophagus or stomach (Project A)
* pts after ER/ESD/RFA for BORN (Project B)
* eradication of BORN and Barrett's esophagus macro- and microscopically (Project B)
* sign agreement with study

Exclusion Criteria:

* macroscopic persistence of Barrett's esophagus (e.g. tongues)
* esophageal varices
* treatment with anticoagulants
* allergy to fluorescein
* polyvalent allergy
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Detection of persistent or recurrent intestinal metaplasia/dysplasia and esophageal and gastric lesions by confocal laser endomicroscopy and classic histopathology | till 3 day after procedure

SECONDARY OUTCOMES:
Sensitivity and specificity of the procedure | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jan Martinek, MD. PhD., Principal Investigator — Institute for Clinical and Experimental Medicine
Locations (1):
- Institute for Clinical and Experimental Medicine, Prague, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Sharma P, Meining AR, Coron E, Lightdale CJ, Wolfsen HC, Bansal A, Bajbouj M, Galmiche JP, Abrams JA, Rastogi A, Gupta N, Michalek JE, Lauwers GY, Wallace MB. Real-time increased detection of neoplastic tissue in Barrett's esophagus with probe-based confocal laser endomicroscopy: final results of an international multicenter, prospective, randomized, controlled trial. Gastrointest Endosc. 2011 Sep;74(3):465-72. doi: 10.1016/j.gie.2011.04.004. Epub 2011 Jul 13. PMID 21741642
- [Background] Meining A, Shah RJ, Slivka A, Pleskow D, Chuttani R, Stevens PD, Becker V, Chen YK. Classification of probe-based confocal laser endomicroscopy findings in pancreaticobiliary strictures. Endoscopy. 2012 Mar;44(3):251-7. doi: 10.1055/s-0031-1291545. Epub 2012 Jan 19. PMID 22261749
- [Background] Shahid MW, Buchner AM, Coron E, Woodward TA, Raimondo M, Dekker E, Fockens P, Wallace MB. Diagnostic accuracy of probe-based confocal laser endomicroscopy in detecting residual colorectal neoplasia after EMR: a prospective study. Gastrointest Endosc. 2012 Mar;75(3):525-33. doi: 10.1016/j.gie.2011.08.024. Epub 2011 Nov 1. PMID 22051243
- [Background] Musquer N, Coquenlorge S, Bourreille A, Aubert P, Matysiak-Budnik T, des Varannes SB, Lauwers G, Neunlist M, Coron E. Probe-based confocal laser endomicroscopy: a new method for quantitative analysis of pit structure in healthy and Crohn's disease patients. Dig Liver Dis. 2013 Jun;45(6):487-92. doi: 10.1016/j.dld.2013.01.018. Epub 2013 Mar 7. PMID 23466186
- [Background] Mannath J, Subramanian V, Kaye PV, Ragunath K. Life-threatening bleeding following Barrett's surveillance biopsies. Endoscopy. 2010;42 Suppl 2:E211-2. doi: 10.1055/s-0030-1255717. Epub 2010 Sep 15. No abstract available. PMID 20845277
- [Background] Kopacova M, Bures J, Osterreicher J, Kvetina J, Pejchal J, Tacheci I, Kunes M, Spelda S, Rejchrt S. Confocal laser endomicroscopy in experimental pigs. Methods of ex vivo imaging. Cas Lek Cesk. 2009;148(6):249-53. PMID 19642306
- [Background] Wang KK, Carr-Locke DL, Singh SK, Neumann H, Bertani H, Galmiche JP, Arsenescu RI, Caillol F, Chang KJ, Chaussade S, Coron E, Costamagna G, Dlugosz A, Ian Gan S, Giovannini M, Gress FG, Haluszka O, Ho KY, Kahaleh M, Konda VJ, Prat F, Shah RJ, Sharma P, Slivka A, Wolfsen HC, Zfass A. Use of probe-based confocal laser endomicroscopy (pCLE) in gastrointestinal applications. A consensus report based on clinical evidence. United European Gastroenterol J. 2015 Jun;3(3):230-54. doi: 10.1177/2050640614566066. PMID 26137298
- [Background] Wallace MB, Crook JE, Saunders M, Lovat L, Coron E, Waxman I, Sharma P, Hwang JH, Banks M, DePreville M, Galmiche JP, Konda V, Diehl NN, Wolfsen HC. Multicenter, randomized, controlled trial of confocal laser endomicroscopy assessment of residual metaplasia after mucosal ablation or resection of GI neoplasia in Barrett's esophagus. Gastrointest Endosc. 2012 Sep;76(3):539-47.e1. doi: 10.1016/j.gie.2012.05.004. Epub 2012 Jun 28. PMID 22749368
- [Background] Konda VJ, Meining A, Jamil LH, Giovannini M, Hwang JH, Wallace MB, Chang KJ, Siddiqui UD, Hart J, Lo SK, Saunders MD, Aslanian HR, Wroblewski K, Waxman I. A pilot study of in vivo identification of pancreatic cystic neoplasms with needle-based confocal laser endomicroscopy under endosonographic guidance. Endoscopy. 2013 Dec;45(12):1006-13. doi: 10.1055/s-0033-1344714. Epub 2013 Oct 25. PMID 24163192
- [Background] Siddiqui AA, Shahid H, Shah A, Khurana T, Huntington W, Ghumman SS, Loren DE, Kowalski TE, Laique S, Hayat U, Eloubeidi MA. High risk of acute pancreatitis after endoscopic ultrasound-guided fine needle aspiration of side branch intraductal papillary mucinous neoplasms. Endosc Ultrasound. 2015 Apr-Jun;4(2):109-14. doi: 10.4103/2303-9027.156728. PMID 26020044
- [Background] Napoleon B, Lemaistre AI, Pujol B, Caillol F, Lucidarme D, Bourdariat R, Morellon-Mialhe B, Fumex F, Lefort C, Lepilliez V, Palazzo L, Monges G, Filoche B, Giovannini M. A novel approach to the diagnosis of pancreatic serous cystadenoma: needle-based confocal laser endomicroscopy. Endoscopy. 2015 Jan;47(1):26-32. doi: 10.1055/s-0034-1390693. Epub 2014 Oct 17. PMID 25325684
- [Derived] Kollar M, Krajciova J, Prefertusova L, Sticova E, Maluskova J, Vackova Z, Martinek J. Probe-based confocal laser endomicroscopy versus biopsies in the diagnostics of oesophageal and gastric lesions: A prospective, pathologist-blinded study. United European Gastroenterol J. 2020 May;8(4):436-443. doi: 10.1177/2050640620904865. Epub 2020 Jan 28. PMID 32213027